CLINICAL TRIAL: NCT04678284
Title: Diabetes Homeless Medication Support Single Arm Treatment Development Trial
Acronym: D-Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HHRI-DHomes; K23DK118117 (NIH)
Record Dates: First submitted 2020-12-17; First posted 2020-12-21 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes; Homeless Persons
Keywords: Type 2 Diabetes; Homeless persons; Delivery of Health Care, Integrated; Primary care; Social determinants of health
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This will be an in-person, phone, or video based behavioral intervention. It will involve a diabetes wellness coach assisting participants to set goals related to diabetes self-care and co-morbidities or social conditions that get in the way of diabetes self-care. There will be encouragement to work on diabetes medication adherence and to address any un/under-treated behavioral health conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D-Homes intervention (Experimental): Behavioral treatments by a diabetes wellness coach as defined below.
  Interventions: Behavioral: Diabetes Homeless Medication Support (D-Homes)

INTERVENTIONS:
Behavioral: Diabetes Homeless Medication Support (D-Homes) — There will be 10 sessions offered within 12 weeks to participants. Sessions will last 30-60 minutes. During sessions a diabetes wellness coach will use behavioral activation and motivational interviewing to get to know participants and set goals to improve diabetes care. The coach will encourage a focus on medication adherence behaviors to the extent that participants are willing. The coach will also help with resource and care coordination. The coach will also provide brief diabetes education as needed.

SUMMARY:
This single-arm trial of the Diabetes Homeless Medication Support intervention alone (n=15) will test the perception and feasibility of anticipated study procedures.

DETAILED DESCRIPTION:
This study is of a set of studies with an overall goal to develop and pilot test a collaborative care intervention using motivational interviewing and behavioral activation alongside education and psychosocial support to improve medication adherence tailored to the experiences of people experiencing homelessness and diabetes (DH). Our team's central hypothesis is that medication adherence and diabetes self-care (and eventual glycemic control, health care use/cost) will improve with an intervention tailored to the unique context of DH.

This protocol addresses a pilot study to test patient perceptions of the feasibility and acceptability of study procedures and refine the D-Homes treatment manual through test cases (n=15). With a hypothesis that the D-Homes manual and study procedures will be feasible and acceptable to DH as measured by self-report and post-treatment interview.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 yrs. or older
2. English-speaking
3. Homelessness by federal definition in the last 12 mo.
4. Self-reported diagnosis of type 2 diabetes, later verified in medical record
5. Plan to stay in local area or be reachable by phone for the next 16 weeks
6. Willingness to work on medication adherence and diabetes self-care
7. HbA1c >/= 7.5%

Exclusion Criteria:

1. Inability to provide informed consent (e.g., presence of a legal guardian, prisoners)
2. Active psychosis or intoxication precluding ability to give informed consent
3. Pregnant or lactating females.
4. Patients who choose to opt out of research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin Healthcare, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
As this work will inform treatment development, we will not share individual participant data. We will submit for publication an overall paper describing our results and how they informed future intervention development.

REFERENCES:
- [Background] Nguyen TD, Attkisson CC, Stegner BL. Assessment of patient satisfaction: development and refinement of a service evaluation questionnaire. Eval Program Plann. 1983;6(3-4):299-313. doi: 10.1016/0149-7189(83)90010-1. PMID 10267258
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Mayberry LS, Gonzalez JS, Wallston KA, Kripalani S, Osborn CY. The ARMS-D out performs the SDSCA, but both are reliable, valid, and predict glycemic control. Diabetes Res Clin Pract. 2013 Nov;102(2):96-104. doi: 10.1016/j.diabres.2013.09.010. Epub 2013 Sep 26. PMID 24209600

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Initial phone screener = 27 In person screen = 23 Excluded = 13 A1c test <7.5% (n = 2) Lost contact (n = 11)
Period: Overall Study
Arm/Group | D-Homes Intervention
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | D-Homes Intervention
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.40 (4.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention
Description: Client Satisfaction Questionnaire, 8-item version, with a score range from 8-32, higher score indicating higher satisfaction.
Time Frame: at 16 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | D-Homes Intervention
Number analyzed (Participants) | 10
score on a scale | 25.4 [17.5 to 33.3]

2. Secondary Outcome: Hemoglobin A1c
Description: Change in point-of-care hemoglobin A1c: This test measures average blood sugar over a three month period, and smaller numbers indicate better glycemic control.
Time Frame: Baseline to 16 weeks
Measure: Mean (95% Confidence Interval); unit: percentage points
Arm/Group | D-Homes Intervention
Number analyzed (Participants) | 10
percentage points | -0.5 [-1.8 to 0.9]

3. Secondary Outcome: Psychological Wellness
Description: Change in psychological wellness as measured by the Short Form (SF)-12. The SF-12 is a self-reported outcome measure assessing psychological wellness and the impact of health on an individual's everyday life. Scores range from 20 to 60, and higher score indicate a higher level of functioning.
Time Frame: Baseline to 16 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | D-Homes Intervention
Number analyzed (Participants) | 10
score on a scale | -2.6 [-14.1 to 8.9]

4. Secondary Outcome: Diabetes Medication Adherence
Description: Change in score on Adherence to Refills and Medications Scales-Diabetes (ARMS-D), Total scores range from 12-48, with higher values indicating worse outcomes.
Time Frame: Baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | D-Homes Intervention
Number analyzed (Participants) | 10
score on a scale | 0.6 [-2.8 to 4.0]

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | D-Homes Intervention
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT04678284/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT04678284/ICF_001.pdf